CLINICAL TRIAL: NCT01480115
Title: A New Tool for Automatic Ovarian Follicle Count and it Abilities to Evaluate Ovarian Reserve
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC11102-11CTLI
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2011-11

CONDITIONS: Infertility
Keywords: antral follicle count; automated antral follicle count; ovarian reserve
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum for FSH, LH, E2, AMH, Prolactin, TSH, Testosterone, Progesterone, 17-OHP, DHEA-S.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: ultrasound examination for AFC evaluation — Ultrasound examination three times during the menstrual cycle to measure the AFC.

SUMMARY:
The ultrasound unit in Meir Medical Center developed new software to automated ovarian follicle count on the basis of 3D US. The investigators intent to evaluate this software at two steps:

* To compared the abilities of the software to physician follicle count.
* To evaluate with the software the antral follicle count, as expression to ovarian reserve at 3 different time of the month.

The investigators believe that the software measurement of the small follicle can be better than the common antral follicle count that is use today, and by this accurate evaluation of the small follicle the investigators can evaluate the ovarian reserve at any time of the mount, and not only at the early follicular phase that use today.

DETAILED DESCRIPTION:
Antral follicle count (AFC) is one of the methods to evaluate ovarian reserve. But this method is not that straightforward with a lot of inter and intra observe variation. In attempt to overcome this problems we going the verified a new software for automated AFC.

At the first step we will compare the human count and the software count of the AFC in 150 exams of ovaries at 3D US.

At the second step we will use the software to evaluate ovarian reserve at 50 women before fertility treatment. This woman will be questioned about epidemiologic data (age, ethnicity, medical history) and evaluate at the early follicular phase with blood test for follicle stimulating hormone, luteinizing hormone , E2, anti-mullerian hormone , Prolactin, thyroid-stimulating hormone, Testosterone, Progesterone, 17-hydroxyprogesterone, dehydroepiandrosterone-Sulphate. The evaluation of the AFC by US will be at early follicular phase, late follicular phase and mid luteal phase

ELIGIBILITY:
Inclusion Criteria:

* woman under age 40 years all
* woman at evaluation before beginning of fertility treatment
* woman with regular menstrual cycle

Exclusion Criteria:

* woman who treat with ovulation induction

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study group will include women faced the fertility unit in Meir Medical Center. Each woman at her first evaluation will invite to volunteer. Also woman during a natural course treatment will invite to volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Antral follicle count accuracy during the menstrual cycle for ovarian reserve evaluation. | Within the 28-35 days of the menstrual cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Tepper, professor, Study Director — Meir Medical Center Israel
Locations (1):
- Fertility unit, Meir Medical Center, Israel, Kfar Saba, Israel

REFERENCES:
- [Background] Hendriks DJ, Mol BW, Bancsi LF, Te Velde ER, Broekmans FJ. Antral follicle count in the prediction of poor ovarian response and pregnancy after in vitro fertilization: a meta-analysis and comparison with basal follicle-stimulating hormone level. Fertil Steril. 2005 Feb;83(2):291-301. doi: 10.1016/j.fertnstert.2004.10.011. PMID 15705365
- [Background] Hendriks DJ, Kwee J, Mol BW, te Velde ER, Broekmans FJ. Ultrasonography as a tool for the prediction of outcome in IVF patients: a comparative meta-analysis of ovarian volume and antral follicle count. Fertil Steril. 2007 Apr;87(4):764-75. doi: 10.1016/j.fertnstert.2006.11.006. Epub 2007 Jan 18. PMID 17239869
- [Background] Raine-Fenning N, Jayaprakasan K, Clewes J. Automated follicle tracking facilitates standardization and may improve work flow. Ultrasound Obstet Gynecol. 2007 Dec;30(7):1015-8. doi: 10.1002/uog.5222. No abstract available. PMID 18044823
- [Background] Styer AK, Toth TL. Antral follicle count in clinical practice: building the bridge from ovarian reserve to in vitro fertilization outcome. Fertil Steril. 2011 Feb;95(2):480-1; discussion 484-5. doi: 10.1016/j.fertnstert.2010.11.054. Epub 2010 Dec 23. PMID 21183169
- [Background] Hsu A, Arny M, Knee AB, Bell C, Cook E, Novak AL, Grow DR. Antral follicle count in clinical practice: analyzing clinical relevance. Fertil Steril. 2011 Feb;95(2):474-9. doi: 10.1016/j.fertnstert.2010.03.023. PMID 20434151
- [Background] Olivennes F, Howies CM, Borini A, Germond M, Trew G, Wikland M, Zegers-Hochschild F, Saunders H, Alam V. Individualizing FSH dose for assisted reproduction using a novel algorithm: the CONSORT study. Reprod Biomed Online. 2011 Feb;22 Suppl 1:S73-82. doi: 10.1016/S1472-6483(11)60012-6. PMID 21575853
- [Background] Al-Azemi M, Killick SR, Duffy S, Pye C, Refaat B, Hill N, Ledger W. Multi-marker assessment of ovarian reserve predicts oocyte yield after ovulation induction. Hum Reprod. 2011 Feb;26(2):414-22. doi: 10.1093/humrep/deq339. Epub 2010 Dec 8. PMID 21147822
- [Background] Deb S, Jayaprakasan K, Campbell BK, Clewes JS, Johnson IR, Raine-Fenning NJ. Intraobserver and interobserver reliability of automated antral follicle counts made using three-dimensional ultrasound and SonoAVC. Ultrasound Obstet Gynecol. 2009 Apr;33(4):477-83. doi: 10.1002/uog.6310. PMID 19212944
- [Background] Murtinger M, Aburumieh A, Rubner P, Eichel V, Zech MH, Zech NH. Improved monitoring of ovarian stimulation using 3D transvaginal ultrasound plus automated volume count. Reprod Biomed Online. 2009 Nov;19(5):695-9. doi: 10.1016/j.rbmo.2009.09.008. PMID 20021717
- [Background] Raine-Fenning N, Jayaprakasan K, Deb S, Clewes J, Joergner I, Dehghani Bonaki S, Johnson I. Automated follicle tracking improves measurement reliability in patients undergoing ovarian stimulation. Reprod Biomed Online. 2009 May;18(5):658-63. doi: 10.1016/s1472-6483(10)60010-7. PMID 19549444